CLINICAL TRIAL: NCT05850520
Title: Randomized, Double-Masked, Active-Controlled, Phase 3 Study of the Efficacy and Safety of Aflibercept 8 mg in Macular Edema Secondary to Retinal Vein Occlusion
Brief Title: A Study to Learn How Well a Higher Amount of Aflibercept Given as an Injection Into the Eye Works and How Safe it is in People With Reduced Vision Due to Swelling in the Macula, Central Part of the Retina Caused by a Blocked Vein in the Retina (Macula Edema Secondary to Retinal Vein Occlusion)
Acronym: QUASAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22153; 2022-502174-16-00 (Other: CTIS (EU))
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Macular Edema Secondary to Retinal Vein Occlusion
MeSH Terms: interventions — aflibercept; salicylhydroxamic acid; Fluorescein Angiography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Higher Dose Regimen 1 (Experimental): Higher dose of aflibercept is administered with initial initiation doses intervals, followed by extension of treatment intervals and further adjustment of intervals according to treatment response.
  Interventions: Drug: Aflibercept, VEGF Trap-Eye(Eylea, BAY86-5321)_higher dose; Drug: Sham; Diagnostic Test: Fluorescein
- Higher Dose Regimen 2 (Experimental): Higher dose of aflibercept is administered with initial initiation doses intervals, followed by extension of treatment intervals and further adjustment of intervals according to treatment response.
  Interventions: Drug: Aflibercept, VEGF Trap-Eye(Eylea, BAY86-5321)_higher dose; Drug: Sham; Diagnostic Test: Fluorescein
- Standard of care (Active Comparator): Aflibercept 2 mg is administered by standard treatment intervals, followed by adjustment of treatment intervals according to treatment response.
  Interventions: Drug: Aflibercept, VEGF Trap-Eye(Eylea, BAY86-5321)_2 mg; Diagnostic Test: Fluorescein

INTERVENTIONS:
Drug: Aflibercept, VEGF Trap-Eye(Eylea, BAY86-5321)_higher dose — Intravitreally (IVT) injection.
  Arms: Higher Dose Regimen 1; Higher Dose Regimen 2
Drug: Aflibercept, VEGF Trap-Eye(Eylea, BAY86-5321)_2 mg — Intravitreally (IVT) injection.
  Arms: Standard of care
Drug: Sham — Sham procedure will be given on visits when an active injection is not planned.
  Arms: Higher Dose Regimen 1; Higher Dose Regimen 2
Diagnostic Test: Fluorescein — Fluorescein 100 mg/mL solution for injection is a dye that makes the retinal vessels visible during FA examinations, and as such, it will be used as an auxiliary medicinal product (AxMP) in this periodic ophthalmic examination. This medicine is for diagnostic use only. It is not used to treat any condition.

SUMMARY:
Researchers are looking for a better way to treat people who have macular edema secondary to retinal vein occlusion (RVO).

In people with RVO, a blood vessel that carries blood away from the retina (vein) becomes blocked. The retina is the very back part of the eye. The blocked vein causes fluid and blood to leak into the retina and thereby causes a swelling of the macula (the center of the retina responsible for fine vision). This swelling is called macular edema.

When a vein in the retina is blocked, the levels of a protein called vascular endothelial growth factor (VEGF) rises. VEGF helps the growth of new blood vessels. This can lead to macular edema and may cause the vision to become blurry.

The study treatment intravitreal (IVT) aflibercept is given as an injection into the eye. It works by blocking VEGF and this can help repair vision problems related to RVO. IVT aflibercept is already available and is prescribed by doctors as the standard of care treatment for macula edema secondary to RVO. Standard of care is a treatment that medical experts consider most appropriate for a disease.

Standard of care is given every 4 weeks in people with macula edema secondary to RVO. While repeated injections of aflibercept may prevent worsening of vision, it may place a burden on the patient. However, a higher amount (8 mg) compared to the standard of care (2 mg) of IVT aflibercept is being tested in studies. This higher amount could be given less often. The amount of IVT aflibercept given is measured in milligrams, also known as mg.

The main purpose of this study is to learn how well a higher amount of the study treatment aflibercept works in people with macular edema secondary to RVO. To answer this, researchers will measure changes in vision called best corrected visual acuity (BCVA) in the study participants between study start and after 36 weeks of treatment. Changes will then be compared between those participants who received the higher amount of IVT aflibercept and those that received standard of care.

To learn how safe the study treatment is in the participants, the researchers will count the number of participants from study start and up to 64 weeks later that have:

* adverse events
* serious adverse events

"Adverse events" are any medical problems that the participants have during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think they might be related to the study treatments. An adverse event is considered "serious" when it leads to death, puts the participants' lives at risk, requires hospitalization, causes disability, causes a baby being born with medical problems or is otherwise medically important.

Dependent on the treatment group, the participants will either receive the higher amount of aflibercept or standard of care as an intravitreal injection for up to 60 weeks. The study will consist of a test (screening) phase, a treatment phase and an end of study phase. Each participant will be in the study for up to 64 weeks.

One visit to the study site is planned during the screening phase, followed by visits approximately every 4 weeks (16 in total) during treatment and one visit at the end of the study.

During the study, the study doctors and their team will:

* check patients' eye health using various eye examination techniques
* measure patients' eye vision (BCVA)
* take blood and urine samples
* do physical examinations
* check vital signs
* examine heart health using electrocardiogram (ECG)
* do pregnancy tests in women of childbearing age

In addition, participants will be asked to fill a questionnaire on vision-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years of age (or country's legal age of adulthood if the legal age is >18 years) at the time of signing the informed consent.
* Treatment-naïve macular edema involving the foveal center secondary to RVO (BRVO, HRVO, or CRVO) diagnosed within 16 weeks (112 days) before the screening visit in the study eye.
* Early Treatment Diabetic Retinopathy Study BCVA letter score of 73 to 24 (20/40 to 20/320) at screening and baseline visits in the study eye.

Decrease in BCVA determined to be primarily the result of RVO in the study eye.

* Mean CST ≥300 μm on optical coherence tomography (OCT) if excluding Bruch's membrane (e.g., Cirrus or Topcon) or ≥320 μm if including Bruch's membrane (e.g., Heidelberg Spectralis), confirmed by the reading center at the screening visit and by the site at baseline visit in the study eye.
* Capable of giving signed informed consent form (ICF) by study participant or legally acceptable representative, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* US participants will be required to have a Health Insurance Portability and Accountability Act (HIPAA) authorization; in other countries, as applicable according to national laws.
* Women of childbearing potential (WOCBP) or men who are sexually active with partners of childbearing potential must agree to use highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 4 months after the last administration of study intervention. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for participation in clinical studies and fulfil the conditions set on Section 10.4.2.

Exclusion Criteria:

* Concurrent disease that causes substantial decrease of BCVA, is expected to limit BCVA recovery or is likely to require medical or surgical intervention during the study in the study eye.
* Presence or history of the following ocular conditions:

  1. Advanced age-related macular degeneration (neovascular AMD or geographic atrophy) in the study eye.
  2. Diabetic macular edema or diabetic retinopathy, defined in diabetic participants as diabetic retinopathy lesions outside the area of the vein occlusion in the study eye and anywhere in the retina in the fellow eye.
  3. Anterior segment neovascularization, vitreous hemorrhage, retinal detachment in the study eye.
  4. Vitreomacular traction, epiretinal membrane or structural damage to the macula that is considered by the Investigator to significantly affect central vision or preclude improvement in vision in the study eye.
  5. Macular hole of stage 2 and above in the study eye.
  6. Myopia of a spherical equivalent of at least 8 diopters prior to any refractive or cataract surgery in the study eye.
  7. Corneal transplant or corneal dystrophy in the study eye.
  8. Idiopathic or autoimmune uveitis in the study or in the fellow eye.
* Presence of the following ocular conditions at screening or baseline visit:

  1. Significant media opacities, including cataract, that interfere with BCVA, or imaging assessments (e.g., fundus photography [FP], OCT) in the study eye.
  2. Aphakia, or pseudophakia with absence of posterior capsule (unless it occurred as a result of a yttrium-aluminum-garnet [YAG] posterior capsulotomy performed more than 30 days before the screening visit), in the study eye.
  3. Uncontrolled glaucoma (defined as IOP >25 mmHg despite treatment with anti-glaucoma medication); or history or likely future need of glaucoma surgery in the study eye.
  4. Intraocular inflammation/infection (including trace, or above, cells in the anterior chamber and/or vitreous) within 12 weeks (84 days) of the screening visit in the study or in the fellow eye.
  5. Extraocular or periocular infection or inflammation (including infectious blepharitis, keratitis, scleritis, or conjunctivitis) in the study or in the fellow eye.
* Uncontrolled blood pressure (defined as systolic >160 mmHg or diastolic >95 mmHg) at the screening visit or baseline visit.
* Uncontrolled diabetes mellitus, defined by hemoglobin A1c (HbA1c) >12% at the screening visit.
* History of cerebrovascular accident or myocardial infarction within 24 weeks (168 days) before the screening visit or between screening and baseline visits.
* Renal failure requiring dialysis, or renal transplant at screening or potentially during the study.
* Any prior or concomitant ocular or systemic treatment (with an investigational or approved, anti-VEGF or other agent) or surgery for RVO in the study eye.
* Previous administration of systemic anti-angiogenic medications for any condition.
* Prior treatment of the study eye with any of the following drugs (any route of ophthalmic administration) or procedures:

  1. Anti-angiogenic drugs at any time including investigational therapy (e.g., with anti-angiopoietin/anti-VEGF bispecific monoclonal antibodies).
  2. Previous use topical steroids within 4 weeks (28 days) from the screening visit, or intraocular or periocular steroids within 16 weeks (112 days) from the screening visit, or steroid implants at any time.
  3. Previous treatment with intraocular or periocular implant, gene therapy, or cell therapy at any time.
  4. Treatment with ocriplasmin at any time.
  5. Vitreoretinal surgery (including scleral buckling) at any time.
  6. Any intraocular surgery, including cataract surgery, within 12 weeks (84 days) before the screening visit.
  7. Previous treatment with retinal laser photocoagulation.
* Prior treatment of the fellow eye with any of the following:

  a. Gene therapy, or cell therapy in the fellow eye at any time.
* Participation in other clinical studies requiring administration of investigational treatments (other than vitamins and minerals) at the time of screening visit, or within 30 days or 5 half-lives of administration of the previous study intervention, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (273):
- United States (53):
  - Retina Consultants of Orange County - Fullerton, Fullerton, California
  - South Coast Retina - Long Beach, Long Beach, California
  - Northern California Retina Vitreous Associates - Mountain View Office, Mountain View, California
  - Desert Retina Consultants - Palm Springs Office, Palm Springs, California
  - Azul Vision Pasadena, Pasadena, California
  - Retina Consultants of Southern California, Redlands, California
  - Retina Consultants of Southern Colorado, PC, Colorado Springs, Colorado
  - New England Retina Associates, New London, Connecticut
  - Rand Eye Institute, Deerfield Beach, Florida
  - National Ophthalmic Research Institute - Fort Myers, Fort Myers, Florida
  - The Eye Institute of West Florida - Largo, Largo, Florida
  - Florida Eye Associates - Melbourne Main Office, Melbourne, Florida
  - Florida Retina Institute - Orlando, Orlando, Florida
  - Retina Specialty Institute - Pensacola, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Associates of Florida - Saint Petersburg, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Center for Retina and Macular Disease - Winter Haven, Winter Haven, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Retina Associates - Elmhurst, Elmhurst, Illinois
  - University Retina and Macula Associates - Oak Forest, Oak Forest, Illinois
  - Retina Associates - Lenexa, Lenexa, Kansas
  - The Retina Care Center - Baltimore, Baltimore, Maryland
  - Cumberland Valley Retina Consultants | Hagerstown, MD, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists - Hagerstown, Hagerstown, Maryland
  - Vitreo-Retinal Associates - Worcester, Grand Rapids, Michigan
  - RCM - St. Louis Park Retina Clinic, Saint Louis Park, Minnesota
  - Retina Consultants of Nevada - Summerlin, Las Vegas, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina - New Brunswick, New Brunswick, New Jersey
  - NJ Retina | Teaneck, Teaneck, New Jersey
  - Vision Research Center, Albuquerque, New Mexico
  - Vitreoretinal Consultants of NY - Great Neck, Great Neck, New York
  - Vitreoretinal Consultants of NY - Hauppauge, Hauppauge, New York
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Retina Associates of Western New York, Rochester, New York
  - Cincinnati Eye Institute - Blue Ash, Blue Ash, Ohio
  - Midwest Retina - Main Office, Dublin, Ohio
  - Retina Consultants, LLC, Salem, Oregon
  - Mid Atlantic Retina - Bethlehem, Bethlehem, Pennsylvania
  - Mid Atlantic Retina - Philadelphia / Wills Eye Hospital, Philadelphia, Pennsylvania
  - Palmetto Retina Center, LLC - Florence, Florence, South Carolina
  - Retina Consultants of South Carolina - Ladson, Ladson, South Carolina
  - Charles Retina Specialists - Germantown, Memphis, Tennessee
  - Austin Retina Associates - Central, Austin, Texas
  - Retina Consultants of Texas - Bellaire, Bellaire, Texas
  - Texas Retina Associates - Fort Worth, Fort Worth, Texas
  - Medical Center Ophthalmology Associates - Northwest, San Antonio, Texas
  - Retina Consultants of Texas - San Antonio Medical Center, San Antonio, Texas
  - Rocky Mountain Retina Consultants - Main Office, Salt Lake City, Utah
  - The Retina Group of Washington - Fairfax, Fairfax, Virginia
  - Spokane Eye Clinical Research - South Hill / Downtown, Spokane, Washington
  - UW Health Carbone Cancer Center, Madison, Wisconsin
- Australia (10):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Marsden Eye Surgery Center, Parramatta, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic, Sydney, New South Wales
  - Sydney West Retina Pty Ltd, Westmead, New South Wales
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Hobart Eye Surgeons, Hobart, Tasmania
  - Centre for Eye Research, East Melbourne, Victoria
  - Lion Eye Institute, Nedlands, Western Australia
- Austria (5):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Medizinische Universität Graz, Graz, Styria
  - Konventhospital Barmherzige Brüder Linz, Linz, Upper Austria
  - Universitätsklinikum AKH Wien, Vienna
  - Hanusch-Krankenhaus Wien, Vienna
- Bulgaria (3):
  - SEHAT Pentagram, Sofia
  - Specialized Hospital For Active Treatment of Eye Diseases Zora, Sofia
  - Spec. Hosp. of Ophthalm. Disease for Active Treatment Varna, Varna
- China (24):
  - The Second Hospital of Anhui medical university, Hefei, Anhui
  - Peking University First Hospital - Oncology Department, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Guangzhou Aier Eye Hospital, Guangzhou, Guangdong
  - Hebei eye hospital, Hebei, Hebei
  - Shijiazhuang General Hospital, Shijiazhuang, Hebei
  - Henan Provincial Eye Hospital, Henan, Henan
  - Tongji Hosp. of Tongji Med Coll, Huazhong Uni of Sci & Tech., Wuhan, Hubei
  - Eye Center of the second Bethune Hospital, jinlin University, Changchun, Jilin
  - The Fourth People's Hospital of Shenyang, Shenyang, Liaoning
  - Aier Eye Hospital (LIAONING), Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region - Opthalmology, Ningxia, Ningxia
  - Shanxi Eye Hospital, Shanxi, Shaanxi
  - Qilu Hosp., Shandong Univ., Jinan, Shandong
  - Aier Eye Hospital (Chengdu), Chengdu, Sichuan
  - ZheJiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Dongyang People's Hospital, Jinhua, Zhejiang
  - Beijing Aier Intech Eye Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Capital Medical University (CMU) - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital CAMS, Beijing
  - Chongqing Aier Ophthalmology Hospital, Chongqing
  - Lanzhou University - The Second Hospital (The Second Clinical Medical College of Lanzhou University), Lanzhou
  - Tianjin Medical University Eye Hospital, Tianjin
- Czechia (7):
  - Fakultní Nemocnice Hradec Kralové, Hradec Králové
  - Fakultní nemocnice Ostrava, Ostrava
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Pardubice
  - Fakultní nemocnice Královské Vinohrady - Urologická klinikay, Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Lexum a.s., Evropska ocni klinika, Prague
  - Axon Clinical, s.r.o., Prague
- Estonia (3):
  - AS Ida-Tallinna Keskhaigla - Oftalmoloogiakeskus, Tallinn
  - Dr. Kai Noor Silmakabinet OÜ, Tallinn
  - Sihtasutus Tartu Ülikooli Kliinikum - Silmakliinik, Tartu
- France (13):
  - Centre Hospitalier National d'Ophthalmologie Quinze-Vingt, Paris, Cedex 12
  - Clinique Rétine Tourny, Bordeaux
  - CHU Bordeaux - Hopital Pellegrin - Ophtalmologie, Bordeaux
  - Hôpital Intercommunal - Créteil Cedex, Créteil
  - CHU Dijon - Hopital Francois Miterrand, Dijon
  - Hôpital de la Croix Rousse, Lyon
  - Centre d'Ophtalmologie - Paradis-Monticelli, Marseille
  - Clinique Jules Verne - Nantes, Nantes
  - Centre d'ophtalmologie de l'Odéon, Paris
  - Centre Ophthalmologie d'Imagerie et de Laser, Paris
  - AP-HP - Hopital Lariboisiere, Paris
  - CM Wolff, Strasbourg
  - Centre Ophtalmologique Transparence - Tours, Tours
- Georgia (2):
  - LTD "IQ Clinic"- Ophthalmology, Tbilisi
  - LTD "Chichua Medical Center MZERA", Tbilisi
- Germany (5):
  - Knappschaftskrankenhaus Sulzbach, Sulzbach, Saarland
  - Uniklinik Bonn / Eye Clinic, Bonn
  - Uni Heidelberg / Augenklinik, Heidelberg
  - Klinikum d. Stadt Ludwigshafen - Ophthalmology, Ludwigshafen
  - St. Franziskus-Hospital Münster - Eye Center, Münster
- Hungary (7):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - University of Semmelweis/ Semmelweis Egyetem, Budapest
  - Budapesti Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Budapest Retina Associates, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Ganglion Medical Center, Pécs
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
- Israel (11):
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Rambam Health Corporation, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center | Internal Medicine Department, Holon
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Centers - HaShalom, Tel Aviv
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (7):
  - Azienda Ospedaliero Universitaria Delle Marche - Clinica Oculistica, Torrette, Ancona
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata - Patologie Retiniche, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oculistica, Rome, Lazio
  - Fondazione G.B.Bietti Per Lo Studio E La Ricerca In Oftalmologia - UOS Retina Medica, Rome, Lazio
  - ASST Fatebenefratelli Sacco, Milan, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Raffaele s.r.l., Milan, Lombardy
- Japan (46):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - University of Fukui Hospital, Yoshida, Fukui
  - Kurume University Hospital, Kurume, Fukuoka
  - Southern Tohoku Eye Clinic, Kōriyama, Fukushima
  - Gunma University Hospital, Maebashi, Gunma
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Kozawa Eye Hospital and Diabetes Center, Mito, Ibaraki
  - Matsumoto Eye Clinic, Toride, Ibaraki
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Medical corporation Eiwakai Dannoue Ophthalmology clinic, Kawasaki, Kanagawa
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Shinshu University Hospital, Matsumoto, Nagano
  - National Defense Medical College Hospital, Tokorozawa, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Shida Eye Clinic, Fujieda-shi, Shizuoka
  - Nihon University Hospital, Chiyoda-ku, Tkyo
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Chofu Eye Clinic, Chōfu, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - Tokyo Metropolitan Institute for Geriatrics and Gerontology, Itabashi-ku, Tokyo
  - Tokiwadai Muranaka Eye Clinic, Itabashi-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Akita University Hospital, Akita
  - Hayashi Eye Hospital, Fukuoka
  - Murakami Karindoh Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kagoshima University Hospital, Kagoshima
  - University of Miyazaki Hospital, Miyazaki
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Okayama University Hospital, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Japanese Red Cross Saitama Hospital, Saitama
  - Toyama University Hospital, Toyama
  - Japanese Red Cross Wakayama Medical Center, Wakayama
  - Yamagata University Hospital, Yamagata
- Latvia (2):
  - Department of Ophthalmology, Riga
  - Riga East Clinical University Hospital "Gailezers", Riga
- Lithuania (2):
  - Hospital of LT University of Health Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (4):
  - Hospital Al-Sultan Abdullah, UiTM | Opthalmology, Bandar Puncak Alam, Selangor
  - Hospital Shah Alam | Ophthalmology, Shah Alam, Selangor
  - Hospital Selayang, Shah Alam, Selangor
  - OasisEye Specialists, Kuala Lumpur
- Poland (9):
  - Prywatna Klinika Okulistyczna OFTALMIKA, Bydgoszcz
  - Specjalistyczny Osrodek Okulistyczny Oculomedica, Bydgoszcz
  - Profesorskie Centrum Okulistyki, Gdansk
  - Gabinet Okulistyczny Prof. Edward Wylegala, Katowice
  - Centrum Medyczne Dietla 19 Sp. z o.o., Krakow
  - Centrum Medyczne PROMED, Krakow
  - Centrum Diagnostyki i Mikrochirurgii Oka Lens, Olsztyn
  - Osrodek Chirurgii Oka prof. Zagorskiego Sp. z o.o., Rzeszów
  - Centrum Medyczne Piasta 47, Wałbrzych
- Portugal (6):
  - AIBILI, Coimbra
  - Espaco Medico de Coimbra, Coimbra
  - CHLC - Hospital dos Capuchos - Servico de Oftalmologia, Lisbon
  - Centro Hospitalar Universitario do Porto, Porto
  - Centro Hospitalar Universitario de Sao Joao | Polo Porto - Centro de Investigacao e Ensaios Clinicos, Porto
  - Centro Hospitalar Vila Nova de Gaia e Espinho | Unit 1 - Clinical Research Center, Porto
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Clinical hospital center Zvezdara, Belgrade
  - Klinicki centar Vojvodine, Novi Sad
- Slovakia (6):
  - Fakultna Nemocnica s poliklinikou F.D.Roosevelta, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Univerzitna nemocnica Bratislava, Nem. Sv. Cyrila a Metoda, Bratislava
  - Fakultna nemocnica Nitra, Nitra
  - Fakultna nemocnica Trencin, Trenčín
  - Specialized hospital for ophthalmology OPHTAL, Zvolen
- South Korea (11):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - University of Ulsan College of Medicine - Asan Medical Center (AMC) - Ophthalmology, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - Samsung Medical Center - Oncology Department, Seoul
  - St. Mary Hospital, Seoul
  - Kim's Eye Hospital, Seoul
- Spain (10):
  - Instituto Oftalmologico Gomez-Ulla S.L. | Oftalmologia, Santiago de Compostela, A Coruña
  - Hospital Universitari General De Catalunya | Oftalmologia, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Puerta De Hierro De Majadahonda | Oftalmologia, Majadahonda, Madrid
  - Hospital Clinic De Barcelona | Oftamologia, Barcelona
  - Hospital Universitari Vall D Hebron | Oftalmologia, Barcelona
  - Hospital De La Santa Creu I Sant Pau | Oftalmologia, Barcelona
  - Clinica Universidad De Navarra | Oftalmologia, Pamplona
  - Hospital General Universitario De Valencia | Oftalmologia, Valencia
  - Hospital Universitario Rio Hortega | Oftalmologia, Valladolid
  - Hospital Universitario Miguel Servet | Oftalmologia, Zaragoza
- Switzerland (5):
  - RétinElysée, Lausanne, Canton of Vaud
  - Inselspital Universitätsspital Bern, Bern
  - Berner Augenklinik am Lindenhofspital, Bern
  - Vista Klinik, Binningen
  - University Eye Hospital Jules Gonin, Lausanne
- Thailand (2):
  - Chiangmai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (7):
  - Ankara Etlik City Hospital | Ophthalmology, Ankara
  - SBU Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Ankara Numune Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Adnan Menderes Universitesi Tip fakultesi, Aydin
  - Ankara Bilkent Sehir Hastanesi, Bilkent Ankara
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
- United Kingdom (10):
  - Hull and East Yorkshire Eye Hospital Hull and East Yorkshire, Hull, East Riding Of Yorkshire
  - Moorfields Eye Hospital, London, Greater London
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - York Teaching Hospital, York, North Yorkshire
  - Frimley Park Hospital NHS, Frimley, Surrey
  - Sunderland Eye Infirmary, Sunderland, Tyne and Wear
  - New Cross Hospital, Wolverhampton, West Midlands
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Leeds Teaching Hospitals NHS Trust | St James's University Hospital - Oncology, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 237 centers in Europe, America, Japan, and Asia-Pacific between 15-May-2023 (first participant first visit) and 07-Nov-2024 (primary completion date).
Pre-assignment Details: In total 1282 participants were screened, of whom 388 participants were screen failures. Overall, 892 participants were randomized and treated. Of these, 838 participants completed the treatment phase through Week 36 (primary completion date).
Groups:
- Aflibercept 2q4: Participants received aflibercept 2 mg administered every 4 weeks.
- Aflibercept 8q8/3: Participants received aflibercept 8 mg administered every 8 weeks, after 3 initial injections at 4-week intervals.
- Aflibercept 8q8/5: Participants received aflibercept 8 mg administered every 8 weeks, after 5 initial injections at 4-week intervals.
Period: Overall Study
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Started | 301 | 293 | 298
Completed (Completed study until Week 36 (primary completion date)) | 287 | 278 | 273
Not Completed | 14 | 15 | 25
Not completed — Withdrawal by Subject | 8 | 8 | 16
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Death | 2 | 2 | 3
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol deviation | 0 | 0 | 1
Not completed — No information was available on whether follow-up was completed or not | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5 | Total
Number analyzed (Participants) | 301 | 293 | 298 | 892
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (11.7) | 65.8 (11.5) | 65.8 (11.5) | 65.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 136 | 146 | 426
  Male | 157 | 157 | 152 | 466
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 25 | 14 | 61
  Not Hispanic or Latino | 267 | 254 | 273 | 794
  Unknown or Not Reported | 12 | 14 | 11 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 2 | 2
  Asian | 101 | 91 | 97 | 289
  Black or African American | 8 | 7 | 9 | 24
  Multiple | 1 | 0 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 1
  Not reported | 13 | 22 | 11 | 46
  White | 178 | 173 | 177 | 528

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA Measured by the ETDRS Letter Score at Week 36
Description: BCVA: Best-Corrected Visual Acuity; ETDRS: Early Treatment Diabetic Retinopathy Study; ETDRS letter score (ranging from 0 to 100 letters). A higher letter score means a better outcome (better visual acuity)
Time Frame: At Week 36
Population: Full analysis set (FAS): All participants randomly assigned to study intervention who were exposed to study intervention (active or sham injection) at least once.
Measure: Least Squares Mean (Standard Error); unit: Letters
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 301 | 293 | 298
Letters | 17.5 (0.7) | 17.4 (0.7) | 18.3 (0.6)
Statistical Analysis 1: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/3; 8q8/3 -2q4; Test type: Non-Inferiority — One-sided test (alpha=0.025) for non-inferiority at a 4-letter margin; p < 0.0001, Mixed Models Analysis — 1-sided p-value; Baseline BCVA measurement was used as a covariate and treatment group, visit, and the stratification variables as fixed factors; Difference in LS means = -0.1, 95% CI 2-sided [-2.0 to 1.9] — Estimation mainly based on hypothetical strategy, i.e. observed data beyond intercurrent events (premature discontinuation of treatment, prohibited medication, missing injection) were censored. Missing/censored data was handled implicitly by MMRM
Statistical Analysis 2: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/5; 8q8/5 -2q4; Test type: Non-Inferiority — One-sided test (alpha=0.025) for non-inferiority at a 4-letter margin; p < 0.0001, Mixed Models Analysis — 1-sided p-value; [statistical method as in outcome 1, analysis 1]; Difference in LS means = 0.8, 95% CI 2-sided [-1.1 to 2.7] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Active Injections From Baseline to Week 36
Description: Active injections refer to the number of injections that were actually administered, as opposed to the number of planned injections.
Time Frame: From baseline to Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of active injections
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 301 | 293 | 298
Number of active injections | 8.8 (0.0) | 6.1 (0.0) | 6.9 (0.0)
Statistical Analysis 1: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/3; 8q8/3 -2q4; Test type: Superiority — Two-sided test (alpha = 0.05); p < 0.0001, ANCOVA — Nominal p-value based on a non-parametric rank ANCOVA adjusted for baseline BCVA, baseline CST, and the stratification variables; Adjusted for baseline BCVA, baseline CST, and the stratification variables; Difference in LS means = -2.7, 95% CI 2-sided [-2.8 to -2.6] — Estimation based on composite strategy for premature treatment discontinuation due to treatment related AEs and hypothetical strategy for premature treatment discontinuation due to other reasons. Hypothetical values imputed using a MI model
Statistical Analysis 2: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/5; 8q8/5 -2q4; Test type: Superiority — Two-sided test (alpha = 0.05); p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Adjusted for baseline BCVA, baseline CST, and the stratification variables; Difference in LS means = -1.8, 95% CI 2-sided [-1.9 to -1.7] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Participants Gaining at Least 15 Letters in BCVA From Baseline at Week 36
Time Frame: From baseline at Week 36
Population: Full analysis set (FAS): All participants randomly assigned and exposed to study intervention (active or sham injection) at least once.
  The Overall Number of Participants Analyzed differs from the Overall Number of Baseline Participants because only observed cases were used, excluding data after an intercurrent event (ICE) (e.g., stopping intervention or using prohibited medication before Week 36). Missing cases were not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 264 | 260 | 248
Participants | 158 | 153 | 161

4. Secondary Outcome: Participants Achieving an ETDRS Letter Score of at Least 69 (Approximate 20/40 Snellen Equivalent) at Week 36
Description: ETDRS letter score (ranging from 0 to 100 letters). A higher letter score means a better outcome (better visual acuity)
Time Frame: At Week 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 264 | 260 | 248
Participants | 179 | 189 | 189

5. Secondary Outcome: Participants Having no Intraretinal Fluid (IRF) and no Sub-retinal Fluid (SRF) in the Center Subfield at Week 36
Description: Number of participants with no retinal fluid (no IRF and no SRF) in the central subfield at Week 36
Time Frame: At Week 36
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 264 | 260 | 247
Participants | 221 | 211 | 202

6. Secondary Outcome: Change From Baseline in Central Sub-field Thickness (CST) at Week 36
Time Frame: From baseline to Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 301 | 293 | 298
μm | -370.8 (3.9) | -370.9 (3.1) | -369.5 (2.3)
Statistical Analysis 1: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/3; 8q8/3 - 2q4; Test type: Superiority — Two-sided test (alpha = 0.05); p = 0.9804, Mixed Models Analysis — Nominal p-value for the two-sided test; Baseline CST measurement was used as a covariate and treatment group, visit, and the stratification variables as fixed factors; Difference in LS means = -0.1, 95% CI 2-sided [-10.0 to 9.8] — Estimation mainly based on hypothetical strategy, i.e. observed data beyond ICE (premature discontinuation of treatment, prohibited medication, missing injection) were censored. Missing/censored data was handled implicitly by MMRM
Statistical Analysis 2: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/5; 8q8/5 - 2q4; Test type: Superiority — Two-sided test (alpha = 0.05); p = 0.7863, Mixed Models Analysis — Nominal p-value for the two-sided test; [statistical method as in outcome 6, analysis 1]; Difference in LS means = 1.2, 95% CI 2-sided [-7.7 to 10.2] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in NEI VFQ 25 Total Score at Week 36
Description: NEI-VFQ-25: National Eye Institute Visual Functioning Questionnaire-25; The NEI VFQ-25 total score ranges from 0 to 100. A higher score means a better outcome (better patient-reported visual function).
Time Frame: From baseline to Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 301 | 293 | 298
Scores on a scale | 6.27 (0.67) | 5.91 (0.61) | 6.92 (0.63)
Statistical Analysis 1: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/3; 8q8/3 - 2q4; Test type: Superiority — Two-sided test (alpha = 0.05); p = 0.6869, ANCOVA — Nominal p-value for the two-sided test; Baseline NEI-VFQ-25 total score measurement used as a covariate and treatment group, visit, and stratification variables as fixed factors; Difference in LS means = -0.36, 95% CI 2-sided [-2.1 to 1.40] — Estimation mainly based on hypothetical strategy, i.e. observed data beyond ICE (premature discontinuation of treatment, prohibited medication, missing active injection) were censored. Missing/censored data was imputed by LOCF approach
Statistical Analysis 2: Comparison: Aflibercept 2q4 vs Aflibercept 8q8/5; 8q8/5 - 2q4; Test type: Superiority; ANCOVA; [statistical method as in outcome 7, analysis 1]; Difference in LS means = 0.65, 95% CI 2-sided [-1.2 to 2.45] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Participants Dosed Only Q8 Through Week 36 in the 8 mg Q8 Group
Description: Number of participants in the aflibercept 8q8/3 and the aflibercept 8q8/5 groups who were able to maintain every 8 weeks (Q8) dosing through Week 36. Only participants who did not discontinue study intervention prior to Week 36, and were therefore considered "completers" for Week 36, were included in the analysis of this endpoint.
Time Frame: Through Week 36
Population: SAF: All participants randomly assigned to study intervention who were exposed to study intervention (active or sham injection) at least once. Analysis of the SAF was performed according to the treatment the participant actually received (as treated).
  The Overall Number of Participants Analyzed is not consistent with numbers provided in the Overall Number of Baseline Participants because only participants considered as completers for Week 36 were included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- All Aflibercept 8 mg: Pooled aflibercept 8 mg administered every 8 weeks, after 3 or 5 initial injections at 4-week intervals.
Arm/Group | Aflibercept 8q8/3 | Aflibercept 8q8/5 | All Aflibercept 8 mg
Number analyzed (Participants) | 278 | 273 | 551
Participants | 246 | 255 | 501

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Through Weeks 36
Description: TEAEs were defined as AEs that occurred in the time frame from first injection (active or sham) to the last injection (active or sham) plus 30 days. Ocular TEAEs in study eye and non-ocular TEAEs are included (ocular TEAEs in fellow eye are excluded)
Time Frame: Through Week 36
Population: Safety analysis set (SAF): All participants randomly assigned to study intervention who were exposed to study intervention (active or sham injection) at least once. Analysis of the SAF was performed according to the treatment the participant actually received (as treated).
Measure: Count of Participants; unit: Participants
Groups:
- All Aflibercept HD: Pooled aflibercept 8 mg administered every 8 weeks, after 3 or 5 initial injections at 4-week intervals.
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5 | All Aflibercept HD
Number analyzed (Participants) | 301 | 293 | 298 | 591
Participants
  Number of participants with TEAEs | 188 | 184 | 176 | 360
  Number of participants with TESAEs | 32 | 23 | 26 | 49

10. Secondary Outcome: Systemic Exposure to Aflibercept as Assessed by Plasma Concentrations of Free, Adjusted Bound and Total Aflibercept From Baseline Through Weeks 36
Description: Total aflibercept is the sum of free and adjusted bound aflibercept.
Time Frame: From baseline through Week 36
Population: Pharmacokinetic analysis set (PKS): All participants randomly assigned to study intervention with at least one non-missing PK result after the first dose of study intervention.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5
Number analyzed (Participants) | 299 | 290 | 294
ng/mL
  Week 4: number analyzed (Participants) | 290 | 279 | 282
  Week 4 | 91.6 (55.82) | 281.8 (52.16) | 270.7 (63.78)
  Week 12: number analyzed (Participants) | 291 | 279 | 276
  Week 12 | 151.5 (56.99) | 451.7 (58.83) | 452.6 (57.04)
  Week 16: number analyzed (Participants) | 272 | 271 | 268
  Week 16 | 241.6 (48.40) | 470.5 (58.24) | 729.0 (43.82)
  Week 24: number analyzed (Participants) | 278 | 265 | 268
  Week 24 | 165.6 (58.72) | 179.8 (73.07) | 202.5 (80.94)
  Week 36: number analyzed (Participants) | 75 | 72 | 75
  Week 36 | 167.8 (58.81) | 366.0 (57.87) | 313.8 (97.30)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the first injection (active or sham) up to the last injection (active or sham) plus 30 days. AE reporting for the all-cause mortality considers all deaths that occurred at any time during the study, up to cut-off date for the primary completion analysis 07 NOV 2024 (approximately 36 weeks).
Description: Ocular treatment-emergent adverse events (TEAEs) in study eye and non-ocular TEAEs (ocular TEAEs in fellow eye are excluded)
Groups:
- Aflibercept 2q4: Participants received aflibercept 2mg administered every 4 weeks.
Arm/Group | Aflibercept 2q4 | Aflibercept 8q8/3 | Aflibercept 8q8/5 | All Aflibercept 8 mg
All-Cause Mortality (participants affected / at risk) | 2/301 | 2/293 | 3/298 | 5/591
Serious Adverse Events (participants affected / at risk) | 32/301 | 23/293 | 26/298 | 49/591
Other Adverse Events (participants affected / at risk) | 188/301 | 184/293 | 176/298 | 360/591
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2q4 (N=301) | Aflibercept 8q8/3 (N=293) | Aflibercept 8q8/5 (N=298) | All Aflibercept 8 mg (N=591)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Primary hyperaldosteronism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vasculitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Macular hole (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Endophthalmitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Medical induction of coma (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2q4 (N=301) | Aflibercept 8q8/3 (N=293) | Aflibercept 8q8/5 (N=298) | All Aflibercept 8 mg (N=591)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Left ventricular enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ventricular dyssynchrony (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thalassaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presbyacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 4 (4) | 6 (6)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphakia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Borderline glaucoma (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 9 (9) | 5 (5) | 9 (9) | 14 (14)
Cataract cortical (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ciliary muscle spasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 6 (7) | 10 (10) | 7 (7) | 17 (17)
Conjunctival irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 4 (5) | 3 (4) | 2 (2) | 5 (6)
Corneal infiltrates (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Corneal scar (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 6 (6) | 4 (4) | 5 (5) | 9 (9)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 3 (3) | 5 (5) | 4 (4) | 9 (9)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 4 (4) | 1 (1) | 5 (5)
Iritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lenticular opacities (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Macular degeneration (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Maculopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 4 (4) | 4 (4) | 2 (2) | 6 (6)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Optic nerve cupping (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 1 (2) | 1 (2) | 1 (1) | 2 (3)
Presbyopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pterygium (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 5 (5) | 4 (5) | 2 (3) | 6 (8)
Retinal artery embolism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Retinal exudates (Eye disorders) | 1 (1) | 2 (2) | 2 (3) | 4 (5)
Retinal haemorrhage (Eye disorders) | 1 (1) | 2 (3) | 2 (2) | 4 (5)
Retinal ischaemia (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Retinal oedema (Eye disorders) | 2 (2) | 2 (2) | 1 (2) | 3 (4)
Retinal pigment epitheliopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Retinal vascular disorder (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Retinal vein occlusion (Eye disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Visual acuity reduced (Eye disorders) | 3 (3) | 12 (12) | 7 (7) | 19 (19)
Visual field defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 2 (2) | 8 (8) | 9 (11) | 17 (19)
Vitreous floaters (Eye disorders) | 3 (4) | 4 (4) | 2 (2) | 6 (6)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Vitreous opacities (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Keratic precipitates (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anterior chamber cell (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Corneal disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anterior chamber disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal drusen (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 6 (6) | 3 (3) | 7 (7) | 10 (10)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular ischaemia (Eye disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Normal tension glaucoma (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Dysmetropsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Narrow anterior chamber angle (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Dry age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal collateral vessels (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Conjunctival suffusion (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Macular thickening (Eye disorders) | 0 (0) | 5 (5) | 0 (0) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (5) | 3 (4) | 7 (9)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (2) | 4 (4) | 1 (1) | 5 (5)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 4 (4) | 0 (0) | 4 (4)
Pain (General disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sensation of foreign body (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Application site hypersensitivity (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (3)
Metabolic dysfunction-associated liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to chemicals (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 4 (4)
Chronic hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (3) | 5 (6)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 6 (6) | 4 (4) | 1 (1) | 5 (5)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (9) | 15 (18) | 14 (15) | 29 (33)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 4 (4)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3) | 3 (4) | 6 (7)
Urinary tract infection (Infections and infestations) | 10 (10) | 4 (4) | 10 (10) | 14 (14)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes dermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 12 (12) | 6 (6) | 18 (18)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 0 (0) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-ocular injection complication (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0) | 5 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood albumin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 5 (6) | 2 (2) | 7 (8)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glucose urine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 2 (2) | 3 (3) | 5 (5) | 8 (8)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 5 (11) | 16 (22) | 15 (25) | 31 (47)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mean cell haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mean cell volume abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
White blood cells urine positive (Investigations) | 1 (1) | 1 (1) | 1 (2) | 2 (3)
Urinary sediment present (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Red blood cells urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Creatinine urine increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Protein urine present (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Urine protein/creatinine ratio increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Creatinine urine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic nerve cup/disc ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Intraocular pressure test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urobilinogen urine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 7 (7) | 10 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 3 (3) | 4 (4)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 4 (4) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 3 (3) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 2 (2) | 5 (6)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0) | 4 (4) | 4 (4)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (14) | 6 (6) | 6 (8) | 12 (14)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infertility (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 2 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 1 (1) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (3)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cutaneous symptom (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Menopause (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 10 (12) | 19 (20) | 20 (22) | 39 (42)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vein disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular shunt (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Brachiocephalic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vein rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scalp haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05850520/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT05850520/SAP_001.pdf